CLINICAL TRIAL: NCT06151938
Title: A Prospective Observational Study Evaluating Relevance of Measurement Instruments in Assessing Effectiveness of ACARIZAX® in the Treatment of Moderate to Severe House Dust Mite Allergic Rhinitis With/Without Allergic Asthma in Chinese
Brief Title: Evaluate Measurement Instruments Relevance in Assessing Effectiveness of ACARIZAX® in House Dust Mite Allergic Rhinitis
Status: Enrolling by invitation | Type: Observational
Sponsor: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NI-MT-08
Record Dates: First submitted 2023-11-16; First posted 2023-11-30 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Allergic Rhinitis Due to House Dust Mite; Allergic Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Standardised allergen extract from house dust mites (ACARIZAX®): Observational study to collect real-world data: patients will be treated with ACARIZAX house dust mite (HDM) sublingual allergy immunotherapy (SLIT) tablet for one tablet per day.
  Interventions: Drug: Standardised allergen extract from house dust mites

INTERVENTIONS:
Drug: Standardised allergen extract from house dust mites — Drug: Allergen immunotherapy [ACARIZAX® (12-SQ HDM) house dust mite (HDM) sublingual allergy immunotherapy (SLIT) tablet] for moderate to severe house dust mite allergic rhinitis with or without allergic asthma for 12 months.
  Other Names: ACARIZAX® (12-SQ HDM)

SUMMARY:
The study is a single-center, observational design with a 12-month duration. Approximately 100 Chinese adult (18-65 years old) and adolescent (12-17 years old) with moderate to severe house dust mite (HDM) allergic rhinitis (AR) with or without allergic asthma (AA) who are newly prescribed ACARIZAX® will be recruited for evaluation of the relevance of measurement instruments. The instruments referred to three patient-report scales of allergic rhinitis symptom and quality-of-life including the Daily symptom score (DSS), Standardised rhinoconjunctivitis quality-of-life questionnaire [RQLQ(S)], and Visual analogue scale (VAS). Other data will be collected to evaluate the effectiveness and safety of ACARIZAX® under real-world clinical practices.

DETAILED DESCRIPTION:
This is a prospective, non-interventional, observational, single-centre, open-label study. Chinese adult (18-65 years old) and adolescent (12-17 years old) HDM AR patients who are newly prescribed with ACARIZAX® at the discretion of attending physician, according to the approved indication by Hainan Provincial Health Commission, will be recruited for this study. Approximately 100 adult (18-65 years old) and adolescent (12-17 years old) patients are expected to be enrolled from Hainan Branch Hospital of Ruijin Hospital. Patients are included in the study only after the decision for treatment with ACARIZAX® has been made, and only with the objective of collecting relevant data about clinical effectiveness and safety of treatment with ACARIZAX® under real-world conditions. No further medical procedures beyond standard care at the discretion of the attending physician are necessary for participation in this study.

Over the 13-month study (including 12-month of treatment), total of 5 scheduled visits will be documented: enrolment and first administration of ACARIZAX® (Visit 1, V0), and subsequent visits performed in 3-month intervals after the first administration at the third month (Visit 2, V1), sixth month (Visit 3, V2), ninth month (Visit 4, V3), and twelfth month (Visit 5, V4) respectively. The actual number and duration of follow-up visits are according to routine practice and may be changed at the physician's discretion. All adverse events (AE) will be collected from the first dose administration until 30 days after the last dose of ACARIZAX® (end of study).

ELIGIBILITY:
Inclusion Criteria:

* Adult and adolescent (12-65 years old) allergic rhinitis patients should meet each of the following criteria:

  * Adult with age of 18-65 years for allergic rhinitis with or without allergic asthma. Adolescent with age of 12-17 years for allergic rhinitis.
  * Clinical history and a positive test of dust mite sensitization (positive skin prick test result ≥+++ or positive specific IgE test result ≥grade 3).
  * Persistent moderate to severe dust mite allergic rhinitis despite use of symptom-relieving medication (symptom assessment defined as to assess symptoms of rhinitis by VAS score≥ 5).
  * Newly prescribed with ACARIZAX®.
  * For adults, must provide signed informed consent; for adolescents, written informed consent must be obtained from both guardian and patient himself/herself if the level of intellectual maturity makes it appropriate.
* Patients with allergic asthma should also meet both of the following criteria:

  * Dust mite induced asthma not well controlled by inhaled corticosteroids and associated with mild to severe dust mite allergic rhinitis.
  * FEV1 ≥ 70% of predicted value after adequate pharmacologic treatment.

Exclusion Criteria:

* Patients with hypersensitivity to any of the excipients.
* Patients with severe asthma exacerbations within the last 3 months.
* Asthmatic patients experiencing an acute respiratory tract infection should have the treatment postponed.
* Patients with acute severe oral inflammation and oral wounds.
* Patients who have previous treatment with Omalizumab within the last 120 days.
* Patient who currently participates in or plan to participate in any interventional clinical study.
* Any other reason that, in the investigator's opinion, makes the patient unsuitable to participate in this study.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients (18-65 years) diagnosed by clinical history and a positive test of house dust mite sensitisation [skin prick test and/or specific Immunoglobulin E (IgE)] with at least one of the following conditions:
  * persistent moderate to severe house dust mite allergic rhinitis despite use of symptom-relieving medication
  * house dust mite allergic asthma not well controlled by inhaled corticosteroids and associated with mild to severe house dust mite allergic rhinitis.
  Adolescents (12-17 years) diagnosed by clinical history and a positive test of house dust mite sensitisation (skin prick test and/or specific IgE) with persistent moderate to severe house dust mite allergic rhinitis despite use of symptom-relieving medication.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-21 (Actual); Primary Completion 2025-05-20 (Estimated); Study Completion 2025-08-20 (Estimated)

PRIMARY OUTCOMES:
Correlation between three measurement instruments | 12 months
  • The correlation between the score changes from baseline to 12 months of treatment (Visit 4) of three measurement instruments (as follows).
  Measurement instruments include:
  * Daily symptom score (DSS) for 7 consecutive days [minimum: 0; maximum: 18; Higher score indicates worse symptoms ]
  * Standardised Rhinoconjunctivitis Quality of Life Questionnaire [RQLQ(S)] score, [minimum: 0; maximum: 168; Higher score indicates worse quality of life]
  * Visual Analog Scale (VAS) value of the global discomfort caused by AR. [minimum: 0mm; maximum: 100mm; Higher score indicates more discomfort caused by AR]

SECONDARY OUTCOMES:
Change in average of Daily Medication Score (DMS) | 12 months
  • The change in average of Daily Medication Score (DMS) for 7 consecutive days from baseline to 12th month of treatment (Visit 4).
  [minimum: 0; maximum: 20; Higher score indicates more medication use]
Change in average of Total Combined Rhinitis Score (TCRS) | 12 months
  • The change in average of Total Combined Rhinitis Score (TCRS) for 7 consecutive days from baseline to 12th month of treatment (Visit 4).
  [TCRS= Rhinitis DSS+ Rhinitis DMS; minimum: 0; maximum: 24; Higher score indicates worse rhinitis symptoms and more rhinitis medication use]
To describe all adverse events (AE) and serious adverse events (SAE) | up to 13 months
  • All AEs and SAEs from the study initiation to the end of study.

OTHER OUTCOMES:
Change in Asthma Control Questionnaire (ACQ) | 12 months
  • Among patients with AR and AA, the change in Asthma Control Questionnaire (ACQ) from baseline to the 12th month of treatment (Visit 4).
  [minimum: 0; maximum: 6; Higher score indicates worse asthma condition]
Change in the Forced Expiratory Volume in One Second (FEV1) | 12 months
  • Among patients with AR and AA, the change in the Forced Expiratory Volume in One Second (FEV1) from baseline to the 12th month of treatment (Visit 4).
Change in the ratio of FEV1 and the Force Vital Capacity (FVC) | 12 months
  • Among patients with AR and AA, the change in the ratio of FEV1 and the Force Vital Capacity (FVC), that is the FEV1/FVC, from baseline to the 12th month of treatment (Visit 4).
Change in the force mid-expiratory flow (FEF25-75%, FEF25%, FEF50%, FEF75%) value | 12 months
  • Among patients with AR and AA, the change in the force mid-expiratory flow (FEF25-75%, FEF25%, FEF50%, FEF75%) value from baseline to the 12th month of treatment (Visit 4).
Change in the Fractional Exhaled Nitric Oxide (FeNO) | 12 months
  • Among patients with AR and AA, the change in the Fractional Exhaled Nitric Oxide (FeNO) from baseline to the 12th month of treatment (Visit 4).
Total AR / (AR with AA) -related treatment costs | 12 months in a 3-month interval.
  To describe the total AR / (AR with AA) - related treatment costs
AR / (AR with AA) -related treatment costs of each outpatient visit, emergency room visit, and hospitalization | 12 months in a 3-month interval
  To describe the AR / (AR with AA) - related treatment costs and break down (if applicable) of each outpatient visit, emergency room visit, and hospitalization
Number of outpatient visit, emergency room visit, and hospitalization due to AR / (AR with AA) | 12 months in a 3-month interval
  To describe the number of outpatient visit, emergency room visit, and hospitalization due to AR / (AR with AA)
Length of stay per hospitalization due to AR / (AR with AA) | 12 months in a 3-month interval
  To describe the length of stay per hospitalization due to AR / (AR with AA)

CONTACTS AND LOCATIONS:
Overall Officials: Wei Tang, PhD, MD, Principal Investigator — Ruijin-Hainan Hospital Shanghai Jiao Tong University School Of Medicine
Locations (1):
- Ruijin-Hainan Hospital Shanghai Jiao Tong University School of Medicine (Hainan Boao Research Hospital), Qionghai, Hainan, China

IPD SHARING:
Plan to Share IPD: No
No sharing plan